CLINICAL TRIAL: NCT02127528
Title: Empiric Antibiotic Therapy for Ventilator-acquired Pneumonia With Gram-negative Bacilli in Intensive Care: Pharmacodynamic Evaluation and Impact.
Brief Title: Empiric Antibiotic Therapy for Ventilator-acquired Pneumonia With Gram-negative Bacilli in Intensive Care
Acronym: TARGET-REA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P1101137
Record Dates: First submitted 2013-11-07; First posted 2014-04-30 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Ventilator-associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
this study aims to verify the adequacy of doses of antibiotics prescribed in clinical practice for the treatment of ventilated acquired pneumonia (VAP) in the intensive care unit (ICU) with the pharmacodynamic efficacy criteria considered relevant literature. The impact of these pharmacodynamic parameters on the clinical and microbiological VAP will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Use of mechanical ventilation for more than 48 hours
2. Clinical suspicion of ventilation-acquired pneumonia (VAP) defined by new radiological persisting infiltrate (or ARDS) AND one of the following features:

   purulent tracheal aspirates OR temperature ≥ 38.3°C OR leukocytosis> 10 giga/L
3. High risk of multidrug-resistant bacteria, defined as either at least 6 days of mechanical ventilation OR antibiotic treatment in the previous 15 days
4. Implementation of a prior distal respiratory sample for microbiological diagnosis by bronchoalveolar lavage (BAL) OR distal sampling by protected catheter (PDP)
5. Age ≥ 18 years
6. Implementing a medical examination
7. Obtain the written consent of the patient, one of its relatives or trusted person previously designated or emergency clause.

Exclusion Criteria:

1. Pregnant woman
2. Expected death within 72 hours of diagnosis of VAP patient
3. Dialysis
4. No affiliation to a social security scheme (beneficiary or legal)
5. Contraindication to one of classes of molecules used antibiotics (β-lactam / Fluoroquinolones / Aminoglycosides), contained in the Summary of Product Characteristics for authorization on the market.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pneumonia acquired in mechanically ventilated patients (PAVM)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
adequate antibiotics | 28 days
  proportion of patients for whom the pharmacodynamic target defined a priori according to data from the literature is reached for each antibiotic anti Gram-negative bacillus used empirically activity (including β-lactams, fluoroquinolones and aminoglycosides)

SECONDARY OUTCOMES:
Bacterial species | 28 days
  Bacterial species in question, defined as any bacteria isolated in significant amounts on the diagnostic breath sampling
Distribution of the main pharmacodynamic parameters | 28 days
  1. ratio of the peak serum level (Cmax) on the minimal inhibitory concentration (MIC), ie Cmax/MIC ratio (for aminoglycosides and fluoroquinolones): distribution in the population and proportion of patients with Cmax/MIC> 10
  2. ratio of the Area Under the serum concentration time Curve (AUC) on the MIC, ie AUC/MIC ratio (for fluoroquinolones) : distribution in the population and proportion of patients with an AUC/MIC ratio> 125
  3. percentage of time spent above the MIC between 2 injections, and trough/MIC ratio (for β-lactams): distribution in the population and proportion of patients with a T>MIC of 100% (intermittent infusion) or trough/MIC> 4 (continuous infusion)
Eradication of gram negative bacilli responsible for VAP | 28 days
  defined as a bacterial count from distal respiratory sample realized during the third day of treatment, less than the threshold for each isolated Gram negative bacilli initially beyond these thresholds
Death | 28 days
Number of days alive without mechanical ventilation | 28 days
Clinical recovery | 28 days
  defined as patient alive with Clinical Pulmonary Infection Score (CPIS) <8
Score of organ failure (SOFA) | 8 days
  repeated measures every 48h for 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- CH Victor Dupouy, Argenteuil, Val d'Oise, France